CLINICAL TRIAL: NCT00375804
Title: Racial Disparity in Prevalence and Survival Rates in Endometrial Cancer
Brief Title: Racial Disparity in Endometrial Cancer
Status: Terminated | Type: Observational
Why Stopped: Funding and logistical difficuties resulted in the withdrawl of the study.
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 357.03
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives for this study:

1. Investigate some of the causes for the racial disparity of endometrial cancer survival rates among black and white women
2. Examine the biologic correlates of aggressive behavior such as estrogen receptor status, p53 and HER-2/neu overexpression, and aromatase activity

DETAILED DESCRIPTION:
Endometrial cancer is the fourth most common cancer among women and the most common gynecologic cancer. Although the incidence of well-differentiated early stage endometrial cancer is higher among white women, there appears to be an increased incidence of aggressive variants with increased mortality rate among blacks.

Reported 5-year survival rate for white women with endometrial cancer is 90% while black women have only 60% survival. (1,2) Black women tend to have more aggressive cancers and more adverse symptoms such as non-endometrioid histology, grade 3 differentiation, and more stage III and IV cancers. (3,7) Many studies have identified and established risk factors and beneficial behaviors for endometrial cancer, most of which are modifiable. Some of the major risks include obesity, hypertension, high fat diet, diabetes, smoking, increased age, hormone replacement therapy, and tamoxifen use. Behaviors associated with decreased risks are use of oral contraceptives, breast feeding, and physical activity. (4)

There is also evidence that biologic factors may contribute to development of malignant endometrial neoplasms. Both mutation and over expression of the p53 tumor suppressor gene is seen in patients with endometrial cancer, especially those in the advanced stages.

Normally, increased levels of p53 are present in cells with damaged DNA. p53 triggers cells to produce more p21, a molecule that binds to cyclin-dependent kinase 2 (Cdk2). In the unbound state, Cdk2 allows cells to progress to the synthesis stage of the cell cycle; therefore, it remains arrested the Gı phase when it is coupled to p21 in an effort to prevent proliferation of abnormal cells. In addition to this mechanism, p53 is thought to be involved in induction of apoptosis. There are indications that black women may exhibit increased incidence of p53 over expression when compared to white women. (5,6,8)

Another biologic factor involved in endometrial cancer is the estrogen receptor. In contrast to p53, presence of estrogen receptors are a positive prognostic factor because they provide a potential avenue for treating endometrial carcinomas. However, the receptors must be functional in order to be advantageous. Some tumors contain mutated estrogen receptors, which cause changes in the metabolic pathway. Individuals with mutated receptors have varying susceptibilities to developing endometrial cancer. (9)

Aromatase is an enzyme involved in converting androgens to estrogens. Both estrogen and aromatase excess has been identified in endometrial cancer, while no aromatase activity has been indicated in the normal endometrium. Most of the aromatase activity appears to be confined to the stromal cells and is correlated with stromal invasion. It may be possible to inhibit aromatase in an effort to decrease estrogen levels and potentially halt cancer growth. (10,11)

Uterine papillary serous carcinoma (UPSC) is an aggressive variant of endometrial cancer characterized by early metastasis, resistance to therapy, and a high mortality rate. Smaller studies suggest that HER-2/neu may be involved in the tumorigenesis of this disease.(13) Overexpression of the HER2/neu receptor in UPSC is an independent variable that is associated with a poorer overall survival, a worse overall prognosis, occurs more frequently in black women, and may contribute to racial disparity in survival. (12,13)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a new case of endometrial carcinoma at the University of Louisville Hospital or in the Norton Healthcare system from 1995-2000

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chart review of subjects diagnosed with endometrial cancer
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2003-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn P. Parker, MD, Principal Investigator — University of Louisville, James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States